CLINICAL TRIAL: NCT04511546
Title: Exploratory Study of BPET, an Investigational Medical Device Without CE-marking for PET Imaging of the Human Brain
Brief Title: Exploratory Study Using a New Head-only PET Scanner
Acronym: ExploreBPET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Positrigo AG (Industry)
Collaborators: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 001
Record Dates: First submitted 2020-08-07; First posted 2020-08-13 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Brain Diseases
MeSH Terms: conditions — Brain Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BPET Scan (Experimental)
  Interventions: Device: BPET Prototype Scan

INTERVENTIONS:
Device: BPET Prototype Scan — Scan on the BPET Prototype PET system and qualitative comparison with a PET image acquired on a conventional clinical PET system.

SUMMARY:
The "BPET prototype" is a small aperture PET scanner. The BPET prototype will be used with patients, which have just finished their regularly scheduled PET examination on a clinical whole body PET system. The radioactive tracer used for this procedure will still be active. This remaining acitivity will be used for an image acquisition with the BPET prototype without the need for an additional radioactive tracer dose.

The control intervention is be a brain PET scan as part of standard clinical routine. It will be done immediately before the scan on the BPET prototype.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving Informed Consent as documented by signature (Appendix Informed Consent Form)
* ability to sit still in the head-only PET scanner for 15 minutes
* Are scheduled to receive a regular brain PET scan as part of clinical routine.
* Male and Female patients 18 years to 80 years of age

Exclusion Criteria:

* Contraindications to PET examination,
* Patient height smaller than 160 cm or taller than 200 cm,
* Patient weight more than 120 kg,
* Patient cannot sit upright for at least 15 minutes,
* Metal implants in the head,
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, severe dementia, etc. of the participant,
* Participation in another study with investigational drug/device within the 30 days preceding and during the present study,
* Previous enrolment into the current study,
* Enrolment of the investigator, his/her family members, employees and other dependent persons.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-10-27 (Actual); Primary Completion 2021-03-05 (Actual); Study Completion 2021-03-05 (Actual)

PRIMARY OUTCOMES:
PET image of the brain | 1 day
  The primary outcome will be a PET image of the brain for each participant taken on BPET. It will be compared against the image taken by the conventional PET machine by a trained physician and judged by whether it could be used for diagnosis and further analysis.

SECONDARY OUTCOMES:
Usability (patient feedback for seat comfort) | 1 day
  The secondary outcome with respect to usability will be feedback from patients with respect to patient seat comfort.
Usability (medical technologist feedback for ease of positioning) | 1 day
  The secondary outcome with respect to usability will be feedback from medical technologist with respect to easiness of patient positioning.

OTHER OUTCOMES:
Assessment of adverse events | During the imaging procedure which should last 15 minutes.
  Safety of the procedure will be assessed by documenting adverse events (description of the adverse events, number of participants)
Assessment of device deficiencies | During the imaging procedure which should last 15 minutes.
  Safety of the procedure will be assessed by documenting device deficiencies (description of the deficiency).
Identification of new risks | During the imaging procedure which should last 15 minutes.
  Safety of the procedure will be assessed by identifying and documenting any new risk.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Hüllner, PD Dr. med., Principal Investigator — University of Zurich
Locations (1):
- PET Center Schlieren, Schlieren, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No